CLINICAL TRIAL: NCT04223921
Title: Therapeutic Optimization in Patients in Acute Geriatric Care at University Hospital of Montpellier: Follow-up One Month After Discharge From Hospital
Brief Title: Therapeutic Optimization in Patients in Acute Geriatric Care at University Hospital of Montpellier
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0581
Record Dates: First submitted 2020-01-02; First posted 2020-01-13 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Geriatrics; Clinical Pharmacy
Keywords: Medication reconciliation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who will be discharged from hospital (acute geriatric: Patients who will be discharged from hospital (acute geriatric care unit) between January and March 2020
  Interventions: Other: Comparison of patient's medicines

INTERVENTIONS:
Other: Comparison of patient's medicines — Comparison of patient's medicines:
  * between patient's discharge from hospital and one month after this discharge (acute geriatric care unit)
  * between patient's admission and discharge from hospital (acute geriatric care unit

SUMMARY:
This study involves patients who will be discharged from Montpellier University Hospital (acute geriatric care unit) between January and March 2020.

The primary objective is to assess the number of difference(s) in patient's medicines between the discharge from hospital (acute geriatric care unit) and one month after this discharge.

The secondary objectives are:

* to assess the number of changes of medicines between the patient's admission and discharge from hospital (acute geriatric care unit);
* to evaluate the number of inappropriate medicines in patient's treatment at hospital admission (in acute geriatric care unit) and one month after the discharge from hospital;
* to evaluate the number of failures found in the transmission of information between the hospital and the general practitioner/pharmacy one month after the patient's discharge from hospital (acute geriatric care unit).

ELIGIBILITY:
Inclusion Criteria:

* patients who will be discharged from hospital (acute geriatric care unit) between January and March 2020 and who will return to their home or to institution for elderly persons
* patients for whom there will be at least one change in their medicines between their admission and their discharge from hospital

Exclusion Criteria:

* Patients who don't want to participate in this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who will be discharged from hospital (acute geriatric care unit) between January and March 2020
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of medicines prescribed | One month after discharge from hospital (acute geriatric care unit)
  Number of medicines prescribed by general practitioner different from those prescribed at patient's discharge from hospital (acute geriatric care unit)

SECONDARY OUTCOMES:
Number of medicines' changes | At patient's discharge from hospital (acute geriatric care unit)
  Number of changes of medicines between the patient's admission and discharge from hospital (acute geriatric care unit)

OTHER OUTCOMES:
Number of inappropriate medicines in patient's treatments | At hospital admission (in acute geriatric care unit)
  Number of inappropriate medicines in patient's treatments at hospital admission (in acute geriatric care unit)
Number of inappropriate medicines in patient's treatments | One month after discharge from hospital (acute geriatric care unit)
  Number of inappropriate medicines in patient's treatments one month after discharge from hospital (acute geriatric care unit)
Number of failures found in the transmission of information between the hospital and the general practitioner/pharmacy | One month after patient's discharge from hospital (acute geriatric care unit)
  Number of failures found in the transmission of information between the hospital and the general practitioner/pharmacy one month after the patient's discharge from hospital (acute geriatric care unit)

CONTACTS AND LOCATIONS:
Overall Officials: DELINGER FAURE, Ph D, Principal Investigator — UH MONTPELLIER
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC